CLINICAL TRIAL: NCT03054571
Title: Correlation Between Somatic Growth and Number of Erupted Deciduous Teeth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Abdallah Ahmed, Cairo,Egypt, Cairo University
Other Study IDs: DAhmed
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Eruption
MeSH Terms: conditions — Exanthema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This investigation seeks to build upon existing evidence that a relationship exists between body mass and timing and the number of erupted teeth.

DETAILED DESCRIPTION:
Alteration in the order of teeth eruption denotes a disorder in normal development of the teeth, rather than delayed or accelerated growth. The more time deviation of teeth eruption from normal, the more possible the presence of a problem in development of teeth. For these reasons having a non-invasive tool such as body mass index to determine if development will be slower than average, could be helpful to the practitioner.

ELIGIBILITY:
Inclusion Criteria:

- Healthy infants aged 5-36 months. 2-Absence of medical and congenital diseases. 3-Full term infants. 4-Residents of Cairo governorate.

Exclusion Criteria:

* Presence of natal and neonatal teeth.

Ages: 5 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be selected according to the following inclusion and exclusion criteria:
  1. Inclusion criteria:
     1. Healthy infants aged 5-36 months.
     2. Absence of medical and congenital diseases.
     3. Full term infants.
     4. Residents of Cairo governorate.
  2. Exclusion criteria:
  Presence of natal and neonatal teeth.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
number of erupted teeth | around 2 months
  the number of erupted erupted teeth will be counted if any part of the tooth appeared

SECONDARY OUTCOMES:
body mass index | around 2 months
  the index will be counted through the equation

IPD SHARING:
Plan to Share IPD: Undecided
publishing through an national journal